CLINICAL TRIAL: NCT06355401
Title: Effect of Maintenance Hormonal Therapy on the Outcome of Patients With DLBCL
Brief Title: Maintenance Hormonal Therapy and DLBCL
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Walaa Gamal Mohamed Soliman, lecturer of clinical oncology, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-Med-24-03--06PD
Record Dates: First submitted 2024-04-04; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: DLBCL; maintenance hormonal therapy; tamoxifen; ERB
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): DLBCL patients who achieve CR
  Interventions: Drug: Tamoxifen 20mg
- group B (No Intervention): DLBCL patients who achieve CR will be under follow up only

INTERVENTIONS:
Drug: Tamoxifen 20mg — maintenance TAM 20 mg daily for DLBCL who achieve CR after chemotherapy and/or radiotherapy and/or BMT
  Arms: group A

SUMMARY:
the study aims to detect the benefit of maintenance tamoxifen after achieving CR with conventional immuno-chemotherapy and/or radiotherapy in patients with DLDCL

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is the most common form of aggressive non-Hodgkin lymphoma. The standard immuno-chemotherapy (R-CHOP) markedly improves the prognosis of DLBCL, but up to 40% of patients still experience relapse or incomplete remission . So, there is a need for new targeted therapy for such malignancy. Recent studies identified a potential novel target in DLBCL, the ESR2 gene, which codes for the estrogen receptor beta (ERβ) protein, a receptor that can be targeted with selective ER modulators (SERMs) such as tamoxifen. Recent data shows that exposure of DLBCL cell lines to tamoxifen (either alone or in combination with CHOP chemotherapy) results in apoptosis and growth inhibition in vitro and in vivo. these data suggest the potential importance of ERβ in the pathogenesis of DLBCL as well as a potential role for tamoxifen in the treatment of DLBCL.50-100 patients with newly diagnosed DLBCL will be treated with standard immuno-chemotherapy according to disease stage with detection of ERB and ERA on the tissue samples using IHC. After the end of chemotherapy treatment patients who achieve CR will be randomized to either receive tamoxifen maintenance (20 mg daily) versus follow up to evaluate possible tamoxifen effect on disease recurrence, DFS and OS.

PT who achieve CR after 2nd line chemotherapy versus post BMT will also be recruited.

ELIGIBILITY:
Inclusion Criteria:

adults 18-75 years old newly diagnosed DLBCL patients who achieve CR after conventional primary treatment can be included PS 0-2

Exclusion Criteria:

less than 18 years or older than 75 years other types of lymphoid neoplasms cardiac comorbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 2-5 years
  the period from CR till 1st relapse
overall survival | 2-5 years
  the period from 1st diagnosis till study end or death

SECONDARY OUTCOMES:
side effects | 2-5 years
  if there is any increase in adverse events while on TAM maintenance